CLINICAL TRIAL: NCT00290771
Title: A Phase II, Open-label, Multicenter Study Evaluating the Efficacy of Imatinib Plus Hydroxyurea (HU) in Patients With Progressive Glioblastoma Multiforme (GBM) Receiving or Not Receiving Enzyme-inducing Anticonvulsant Drugs (EIACDs)
Brief Title: Efficacy and Safety of Imatinib Mesylate Plus Hydroxyurea (HU) in Patients With Recurrent Glioblastoma Multiforme (GBM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571H2201; CSTI571H2202 (Other: Novartis Pharmaceuticals); NCT00292149 (obsolete NCT alias)
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2011-05-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-04

CONDITIONS: Recurrent Glioblastoma Multiforme (GBM)
Keywords: imatinib mesylate; hydroxyurea; protein tyrosine kinases; glioma; glioblastoma multiforme; recurrent glioblastoma multiforme; GBM; MacDonald criteria
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Imatinib Mesylate; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imatinib 600 mg + hydroxyurea 1000 mg (Experimental): Patients took imatinib 600 mg (1 imatinib 400 mg tablet and 2 imatinib 100 mg tablets) orally once daily with the morning meal. Patients were instructed to swallow the tablets while drinking a large glass of water. In addition to imatinib, patients took hydroxyurea 500 mg orally twice daily with the morning and evening meals. Patients were not allowed concomitant use of enzyme-inducing anticonvulsant drugs.
  Interventions: Drug: Imatinib tablets; Drug: Hydroxyurea capsules
- Imatinib 1000 mg + hydroxyurea 1000 mg (Experimental): Patients took imatinib 500 mg (1 imatinib 400 mg tablet and 1 imatinib 100 mg tablet) orally twice daily with the morning and evening meals. Patients were instructed to swallow the tablets while drinking a large glass of water. In addition to imatinib, patients took hydroxyurea 500 mg orally twice daily with the morning and evening meals. Patients were allowed concomitant use of enzyme-inducing anticonvulsant drugs.
  Interventions: Drug: Imatinib tablets; Drug: Hydroxyurea capsules

INTERVENTIONS:
Drug: Imatinib tablets — Imatinib was supplied as 100 and 400 mg tablets by Novartis.
  Other Names: Glivec®
Drug: Hydroxyurea capsules — Hydroxyurea was supplied locally as 500 mg capsules.

SUMMARY:
This was an investigational study to assess the objective overall response (OOR) rate (complete response [CR] + partial response [PR]) of imatinib mesylate and hydroxyurea (hydroxycarbamide) combination therapy in patients with recurrent glioblastoma multiforme (brain tumors). This study also evaluated the duration of tumor response (as per MacDonald criteria), clinical benefit, progression-free survival rate at 6 and 12 months, and the survival rate at 12 and 24 months.

DETAILED DESCRIPTION:
This ClinicalTrials.gov record includes the results from two studies (Novartis protocol IDs CSTI571H2201 and CSTI571H2202) which were conducted separately but reported together in a single clinical study report. Both studies were phase II, open-label, multicenter, single-arm studies that evaluated the efficacy of imatinib mesylate plus hydroxyurea in subjects with progressive glioblastoma multiforme. The studies were identical in design with two exceptions: Patients in study CSTI571H2201 received a dose of imatinib 600 mg once daily and were not allowed concomitant use of enzyme-inducing anticonvulsant drugs (EIACDs); patients in study CSTI571H2202 received a dose of imatinib 500 mg twice daily and were allowed concomitant use of EIACDs.

ELIGIBILITY:
Inclusion criteria:

* Males and females ≥ 18 years old.
* Histologically-confirmed diagnosis of progressive primary glioblastoma multiforme (GBM) based on original diagnosis. Patients with prior low-grade glioma were eligible if histological re-assessment demonstrated transformation to GBM.
* No more than one prior episode of progressive disease following previously received surgery and/or radiation and only one prior chemotherapy exposure of either temozolomide (TMZ) or nitrosourea including the application of polifeprosan (Gliadel®) wafers.
* Presence of measurable disease on gadolinium-enhanced magnetic resonance imaging (MRI).
* Patients taking steroids must have been on a stable dose for ≥ 7 days.
* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2.
* Hemoglobin ≥ 10 g/dL (or hematocrit > 29%), absolute neutrophil count (ANC) > 1500 cells/L, platelets > 100,000 cells/L.
* Serum creatinine < 1.5 mg/dL, blood urea nitrogen (BUN) < 25 mg/dL, serum aspartate aminotransferase (AST) and bilirubin < 1.5 x upper limit of normal (ULN).
* Sexually-active male and female patients were required to use double-barrier contraception (oral contraceptive plus barrier contraceptive) or must have undergone clinically documented total hysterectomy, ovariectomy, or tubal ligation.
* Female patients of childbearing potential must have had a negative pregnancy test within 48 hours prior to start of study drug.
* Life expectancy ≥ 8 weeks.
* Signed informed consent by the patient prior to patient entry and any study procedure.

Exclusion Criteria:

* Receipt of imatinib or hydroxyurea (HU) prior to study entry or receipt of any investigational agent within the last 6 months.
* Patients who had received a second course of chemotherapy or radiotherapy, unless given as a single localized application of radio surgery.
* In study STI571H2201 only, receipt of enzyme-inducing anticonvulsant drugs (EIACDs), eg, carbamazepine, phenobarbital, phenytoin, fosphenytoin, oxcarbazepine, or primidone. Previous EIACD should have been interrupted 4 weeks prior to study start.
* Grade ≥ 2 peripheral edema or pulmonary or pericardial effusions or ascites of any grade.
* Presence of any uncontrolled systemic infection.
* Patients who were not a minimum of 12 weeks from completion of conventional external beam radiotherapy unless:

  1. There was new radiographical enhancement outside the field of radiation, or
  2. There was new pathological confirmation of recurrent tumor, or
  3. Progressive radiographical enhancement noted on post-radiotherapy/TMZ continue to worsen after an additional course of TMZ.
* Evidence of intra-tumor hemorrhage on pretreatment diagnostic imaging, except for stable post-operative Grade 1 hemorrhage, patients with an excessive risk of an intracranial hemorrhagic event, and patients with history of central nervous system (excluding post-operative Grade 1) or intraocular bleed.
* Patients who had undergone major surgery within 2 weeks prior to study entry or who had not recovered from prior major surgery, patients who had received chemotherapy within 4 weeks prior to study start, or who have not recovered from toxic effects of such therapy.
* Impairment of gastrointestinal function or gastrointestinal disease that could significantly alter the absorption of imatinib.
* Patients taking warfarin sodium.
* Known history of human immunodeficiency virus (HIV) seropositivity; testing for HIV was not required at study entry.
* For the purposes of MRI, patients with a pacemaker, ferromagnetic metal implants other than those approved as safe for use in MR scanners (eg, some types of aneurysm clips, shrapnel), patients suffering from uncontrollable claustrophobia, or those physically unable to fit into the machine (eg, obesity).
* Patients considered by the investigator as unlikely to be compliant with the study, take the study medications, travel for the necessary assessment visits, or have other medical conditions likely to interfere with the study assessments.
* Patients with another primary malignancy treated within the prior 3 years except excised squamous cell carcinomas of the skin and carcinoma in situ lesions of other organs which had been treated for cure.
* Patients not able to provide reliable informed consent and who did not have a legal representative for healthcare decisions on their behalf.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2006-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Reardon, Dr., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg
Started | 131 | 100
Completed | 4 | 3
Not Completed | 127 | 97
Not completed — Disease progression | 95 | 73
Not completed — Death | 11 | 10
Not completed — Adverse Event | 12 | 6
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Administrative problems | 2 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg | Total
Number analyzed (Participants) | 131 | 100 | 231
Age Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.9) | 52.8 (11.4) | 53.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 35 | 87
  Male | 79 | 65 | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an Objective Overall Response (OOR)
Description: Patients with an OOR were those whose best response to treatment was a complete response (CR) or a partial response (PR) assessed with magnetic resonance imaging. A patient had a CR if the target tumors disappeared. A patient had a PR if there was a ≥ 50% reduction in the sum of the products of the largest perpendicular diameters of the target tumors compared to the baseline value. A best response of CR required at least 2 determinations of CR at least 4 weeks apart. A best response of PR required at least 2 determinations of PR or better at least 4 weeks apart (and not qualifying for CR).
Time Frame: Baseline to end of study (Month 24)
Population: Intent-to-treat (ITT) population: All patients who received at least 1 dose of any of the 2 study drugs.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Patients - Imatinib 600 or 1000 mg + Hydroxyurea 1000 mg: Patients took either imatinib 600 mg (1 imatinib 400 mg tablet and 2 imatinib 100 mg tablets) orally once daily with the morning meal or imatinib 500 mg (1 imatinib 400 mg tablet and 1 imatinib 100 mg tablet) orally twice daily with the morning and evening meals. Patients were instructed to swallow the tablets while drinking a large glass of water. In addition to imatinib, patients took hydroxyurea 500 mg orally twice daily with the morning and evening meals.
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg | All Patients - Imatinib 600 or 1000 mg + Hydroxyurea 1000 mg
Number analyzed (Participants) | 131 | 100 | 231
Percentage of participants | 3.8 [1.3 to 8.7] | 3.0 [0.6 to 8.5] | 3.5 [1.5 to 6.7]

2. Secondary Outcome: Duration of Objective Overall Response (OOR)
Description: Duration of OOR only included patients whose best overall response was complete response (CR) or partial response (PR). The start date was the date of the first documented response (CR or PR); the end date was the date of the first documented disease progression (PD) or death from any cause. (PD) was defined as ≥ 25% increase in size of the sum of the products of the largest perpendicular diameters of the target tumors compared to the smallest value recorded at or after baseline. If a patient had not progressed or died, the duration of OOR was censored at the time of the last OOR assessment.
Time Frame: Baseline to end of study (Month 24)
Population: Intent-to-treat (ITT) population: All patients who received at least 1 dose of any of the 2 study drugs.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg | All Patients - Imatinib 600 or 1000 mg + Hydroxyurea 1000 mg
Number analyzed (Participants) | 131 | 100 | 231
Weeks | 41.1 [32.1 to 53.6] | 32.1 [20.1 to NA] — The upper bound of the confidence interval was non-estimable. | 37.1 [32.1 to 53.6]

3. Secondary Outcome: Percentage of Patients Who Had Clinical Benefit
Description: Patients who had clinical benefit were patients with a best response of complete response (CR), partial response (PR), or stable disease (SD) lasting for more than 6 months from the start of treatment until the first documented disease progression (PD) or death from any cause. (PD) was defined as ≥ 25% increase in size of the sum of the products of the largest perpendicular diameters of the target tumors compared to the smallest value recorded at or after baseline. SD was defined as insufficient tumor shrinkage to qualify for PR or CR and no increase in lesions which would qualify as PD.
Time Frame: Baseline to end of study (Month 24)
Population: Intent-to-treat (ITT) population: All patients who received at least 1 dose of any of the 2 study drugs.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg | All Patients - Imatinib 600 or 1000 mg + Hydroxyurea 1000 mg
Number analyzed (Participants) | 131 | 100 | 231
Percentage of participants | 9.9 [5.4 to 16.4] | 6.0 [2.2 to 12.6] | 8.2 [5.0 to 12.5]

4. Secondary Outcome: Percentage of Patients With Progression-free Survival at Months 6 and 12
Description: Progression-free survival (PFS) was defined as the time from the start of treatment to the date of the first documented disease progression (PD) or death due to any cause. (PD) was defined as ≥ 25% increase in size of the sum of the products of the largest perpendicular diameters of the target tumors compared to the smallest value recorded at or after baseline. If a patient had not progressed or died, progression-free survival was censored at the time of the last overall response assessment.
Time Frame: Months 6 and 12
Population: Intent-to-treat (ITT) population: All patients who received at least 1 dose of any of the 2 study drugs.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg | All Patients - Imatinib 600 or 1000 mg + Hydroxyurea 1000 mg
Number analyzed (Participants) | 131 | 100 | 231
Percentage of participants
  6 Months | 11.2 [5.7 to 16.6] | 9.9 [3.8 to 15.9] | 10.6 [6.5 to 14.7]
  12 Months | 6.9 [2.4 to 11.3] | 3.3 [0.0 to 6.9] | 5.3 [2.3 to 8.3]

5. Secondary Outcome: Percentage of Patients Surviving at Months 6, 12, and 24
Description: Patients not known to have died were censored at the time of last survival follow-up.
Time Frame: Months 6, 12, and 24
Population: Intent-to-treat (ITT) population: All patients who received at least 1 dose of any of the 2 study drugs.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg | All Patients - Imatinib 600 or 1000 mg + Hydroxyurea 1000 mg
Number analyzed (Participants) | 131 | 100 | 231
Percentage of participants
  6 Months | 49.2 [40.7 to 57.8] | 50.9 [40.9 to 61.0] | 50.0 [43.4 to 56.5]
  12 Months | 28.5 [20.7 to 36.2] | 31.3 [21.9 to 40.7] | 29.7 [23.7 to 35.7]
  24 Months | 10.7 [3.3 to 18.1] | 20.3 [11.8 to 28.9] | 13.9 [8.0 to 19.7]

6. Secondary Outcome: Number of Patients With at Least 1 Adverse Event
Description: An adverse event (AE) is any undesirable sign, symptom, or medical condition occurring after starting study drug even if the event is not considered to be related to study drug. Study drug refers to imatinib or hydroxyurea. The study treatment is the combination of these two study drugs.
Time Frame: Baseline to end of study (Month 24)
Population: Safety population: All patients who received at least 1 dose of either of the 2 study drugs and who had at least 1 post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg | All Patients - Imatinib 600 or 1000 mg + Hydroxyurea 1000 mg
Number analyzed (Participants) | 131 | 100 | 231
Participants | 129 | 98 | 227

ADVERSE EVENTS:
Description: The analysis was done on the safety population which consisted of 131 patients in the imatinib 600 mg plus hydroxyurea 1000 mg group and 99 patients in the imatinib 1000 mg plus hydroxyurea 1000 mg group.
Arm/Group | Imatinib 600 mg + Hydroxyurea 1000 mg | Imatinib 1000 mg + Hydroxyurea 1000 mg
Serious Adverse Events (participants affected / at risk) | 62/131 | 53/99
Other Adverse Events (participants affected / at risk) | 122/131 | 95/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib 600 mg + Hydroxyurea 1000 mg (N=131) | Imatinib 1000 mg + Hydroxyurea 1000 mg (N=99)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Amaurosis (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Palatal oedema (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 5
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 10 | 3
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 2
Sudden death (General disorders) | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic embolus (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Blood amylase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 12
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 2 | 2
Ataxia (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 2
Cerebral cyst (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 6 | 5
Depressed level of consciousness (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 3
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 4
Hemiparesis (Nervous system disorders) | 2 | 3
Hemiplegia (Nervous system disorders) | 2 | 2
Hypokinesia (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 4 | 4
Loss of consciousness (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 3 | 1
Tongue biting (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 4
Disorientation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Personality change due to a general medical condition (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Staring (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 2 | 2
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib 600 mg + Hydroxyurea 1000 mg (N=131) | Imatinib 1000 mg + Hydroxyurea 1000 mg (N=99)
Anaemia (Blood and lymphatic system disorders) | 19 | 10
Leukopenia (Blood and lymphatic system disorders) | 8 | 9
Lymphopenia (Blood and lymphatic system disorders) | 3 | 7
Neutropenia (Blood and lymphatic system disorders) | 15 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 10
Cushingoid (Endocrine disorders) | 5 | 8
Eyelid oedema (Eye disorders) | 17 | 8
Vision blurred (Eye disorders) | 8 | 5
Constipation (Gastrointestinal disorders) | 22 | 9
Diarrhoea (Gastrointestinal disorders) | 27 | 16
Nausea (Gastrointestinal disorders) | 49 | 37
Vomiting (Gastrointestinal disorders) | 40 | 22
Asthenia (General disorders) | 15 | 13
Face oedema (General disorders) | 7 | 6
Fatigue (General disorders) | 40 | 37
General physical health deterioration (General disorders) | 8 | 7
Oedema (General disorders) | 12 | 1
Oedema peripheral (General disorders) | 31 | 24
Pain (General disorders) | 7 | 1
Pyrexia (General disorders) | 7 | 7
Nasopharyngitis (Infections and infestations) | 10 | 8
Oral candidiasis (Infections and infestations) | 6 | 6
Urinary tract infection (Infections and infestations) | 8 | 4
Anorexia (Metabolism and nutrition disorders) | 10 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 7
Amnesia (Nervous system disorders) | 7 | 8
Aphasia (Nervous system disorders) | 4 | 7
Ataxia (Nervous system disorders) | 11 | 11
Balance disorder (Nervous system disorders) | 0 | 5
Cognitive disorder (Nervous system disorders) | 10 | 13
Convulsion (Nervous system disorders) | 7 | 2
Dizziness (Nervous system disorders) | 13 | 15
Epilepsy (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 33 | 20
Hemiparesis (Nervous system disorders) | 6 | 7
Peripheral motor neuropathy (Nervous system disorders) | 15 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 6
Somnolence (Nervous system disorders) | 12 | 7
Speech disorder (Nervous system disorders) | 8 | 8
Tremor (Nervous system disorders) | 10 | 7
Confusional state (Psychiatric disorders) | 16 | 11
Insomnia (Psychiatric disorders) | 15 | 9
Mood altered (Psychiatric disorders) | 8 | 6
Incontinence (Renal and urinary disorders) | 4 | 5
Sexual dysfunction (Reproductive system and breast disorders) | 7 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Petechiae (Skin and subcutaneous tissue disorders) | 10 | 7
Rash (Skin and subcutaneous tissue disorders) | 14 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.